CLINICAL TRIAL: NCT06545162
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation, Phase I Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of CPX101 in Healthy Volunteers and Overweight or Obese Patients With Multiple Doses
Brief Title: Safety, Tolerability, and Pharmacokinetics of a Single or Multiple Ascending Doses of CPX101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Chia Tai Innovative Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPX101-I-01
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity
Keywords: GLP-1R
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Experimental)
  Interventions: Biological: CPX101 or placebo 80mg single dose
- SAD Cohort 2 (Experimental)
  Interventions: Biological: CPX101 or placebo 120mg single dose
- SAD Cohort 3 (Experimental)
  Interventions: Biological: CPX101 or placebo 160mg single dose
- MAD Cohort 1 (Experimental)
  Interventions: Biological: CPX101 or placebo 80mg Q2W
- MAD Cohort 2 (Experimental)
  Interventions: Biological: CPX101 or placebo 120mg Q2W
- MAD Cohort 3 (Experimental)
  Interventions: Biological: CPX101 or placebo 160mg Q2W
- MAD Cohort 4 (Experimental)
  Interventions: Biological: CPX101 or placebo 200mg Q2W
- SAD cohort 4 (Experimental): 200mg
  Interventions: Biological: CPX101 or placebo 200mg single dose

INTERVENTIONS:
Biological: CPX101 or placebo 80mg single dose — Subcutaneous injection of CPX101 or placebo
  Arms: SAD Cohort 1
Biological: CPX101 or placebo 120mg single dose — Subcutaneous injection of CPX101 or placebo
  Arms: SAD Cohort 2
Biological: CPX101 or placebo 160mg single dose — Subcutaneous injection of CPX101 or placebo
  Arms: SAD Cohort 3
Biological: CPX101 or placebo 80mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: MAD Cohort 1
Biological: CPX101 or placebo 120mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: MAD Cohort 2
Biological: CPX101 or placebo 160mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: MAD Cohort 3
Biological: CPX101 or placebo 200mg Q2W — Subcutaneous injection of CPX101 or placebo
  Arms: MAD Cohort 4
Biological: CPX101 or placebo 200mg single dose — CPX101 or placebo 200mg single dose
  Arms: SAD cohort 4

SUMMARY:
This randomized, double-blind, placebo-controlled Phase I clinical study was designed to evaluate the tolerability and safety, PK profile, immunogenicity of CPX101 in a single dose in healthy participants and multiple doses in overweight and obese patients, and to initially explore the efficacy of multiple doses in weight loss. The study was divided into two parts: single administration and dose escalation (SAD) and multiple administration and dose escalation (MAD).

DETAILED DESCRIPTION:
SAD: Three dose levels (80mg, 120mg, 160mg and200mg) were preset for this phase, and a total of 32 healthy participants were planned to be included. According to the dose increment principle, starting from the dose of 80mg, increasing successively to the high dose, and proceeding in sequence.

MAD: The study was planned to include 48 adult overweight or obese participants, with a preset group of four cohorts, each with 12 participants. MAD1 to MAD 3cohorts were dosed with titration starting at 40mg and given once 1 week (QW) in each cohort. Up to the target dose of 80mgQ2W, 120mg Q2W and 160mg Q2W whereas MAD4 cohort were dosed with titration starting at 80mg and gived once 2week (Q2W) and up to target dose of 240 mg and exploratory of 320mg

ELIGIBILITY:
Inclusion Criteria:

SAD inclusion criteria:

1. Healthy male or female participants aged 18 to 65 (inclusive) at the time of signing the informed consent form;
2. When screening, body mass index (BMI)>20 and<28 kg/m2;
3. During the entire study period, participants must agree to maintain stable dietary and physical activity habits, and have no plans to change their dietary or exercise habits or lose weight;
4. Participants are able to understand and voluntarily sign a written Informed Consent Form (ICF), and are able to complete the relevant procedures and checks in accordance with the protocol;
5. Female participants must meet the following conditions:

   1. No possibility of reproduction;
   2. Possible fertility: The serum pregnancy test result was negative during screening, and effective contraceptive measures were agreed to be taken throughout the entire trial period and within 12 weeks after the last dose. Egg donation is not allowed within 12 weeks after the last dose;
6. Male participants whose female partners have the potential to conceive must take effective contraceptive measures throughout the entire trial period and within 12 weeks after the last dose, and are not allowed to donate sperm.

MAD inclusion criteria:

1. Male or female participants aged 18 to 75 (inclusive) at the time of signing the informed consent form;
2. When screening, obese individuals with 28 ≤ BMI<40kg/m2, or overweight individuals with 24 ≤ BMI<28kg/m2 and at least one of the following weight related comorbidities;
3. During the first 3 months of screening, the weight remained stable;
4. Willing to maintain a stable diet and exercise habits according to the research protocol throughout the entire study period;
5. Participants are able to understand and voluntarily sign a written informed consent form (ICF), and are able to complete the relevant procedures and checks in accordance with the protocol;
6. Female participants must meet the following conditions:

   1. No possibility of reproduction;
   2. Possible fertility: The serum pregnancy test result was negative during screening, and effective contraceptive measures were agreed to be taken throughout the entire trial period and within 12 weeks after the last dose. Egg donation is not allowed within 12 weeks after the last dose;
7. Male participants whose female partners have the potential to conceive must take effective contraceptive measures throughout the entire trial period and within 12 weeks after the last dose, and are not allowed to donate sperm.

Exclusion Criteria:

SAD exclusion criteria:

1. When screening, if there is a medical history or clinical evidence showing that participants have obvious accompanying diseases (including but not limited to cardiovascular, respiratory, digestive, urinary, neurological/psychiatric, blood, immune, endocrine and metabolic, infection, etc.);
2. During the screening period, acute diseases with clinical significance (such as gastrointestinal diseases, gallbladder diseases, pancreatitis), infections (such as influenza, upper respiratory tract infections), which are judged by the investigator to be not suitable for participants in the trial;
3. Use any prescription medication (excluding hormonal contraceptives), over-the-counter medication, herbal medicine, or health supplement within the first 30 days of randomization;
4. When screening, the physical examination or laboratory test results meet any of the following criteria:

   1. Resting systolic blood pressure (SBP)>140mmHg or<90mmHg, and/or diastolic blood pressure (DBP)>90mmHg or<60mmHg (allow retesting after 10 minutes);
   2. When screening, the heart rate should be greater than 100 beats per minute or less than 50 beats per minute (allowing for retesting after 10 minutes);
   3. Hepatic dysfunction;
   4. Renal dysfunction;
   5. During screening, the QTc of ECG examination abnormal;
   6. Positive results in urine drug screening or alcohol breath test during screening;
   7. When screening, hepatitis B surface antigen (HBsAg) is positive, or syphilis antibody is positive, or human immunodeficiency virus (HIV) antibody is positive, or hepatitis C virus (HCV) antibody is positive;
   8. During screening, hemoglobin levels abnormal;
   9. Calcitonin ≥ 20ng/L;
   10. Glycated hemoglobin ≥ 6.5%;
   11. Thyroid dysfunction;
   12. Positive serum pregnancy test during screening;
5. History or family history of medullary thyroid carcinoma, multiple endocrine tumors (MEN) 2A or 2B syndrome;
6. Screening for any type of malignant tumor (whether cured or not) within the previous 5 years, except for locally cured basal cell carcinoma of the skin;
7. Had weight loss surgery (except acupuncture and moxibustion weight loss and local liposuction) within 1 year before screening, or planned to have any weight loss surgery or receive other weight loss treatment during the study period;
8. The Investigator determines the subject who has a history of severe trauma, infection, or major surgery within the past month prior to screening are not suitable to participate in this study;
9. Screening for individuals with a history of drug abuse or drug dependence within the previous year;
10. Have a history of alcohol abuse within the year before screening, or frequently drink alcohol within the 6 months before screening;
11. Screening for individuals who have used any clinical trial drug or are currently undergoing other clinical trials within the previous 3 months, or whose trial drug is still within 5 half-lives (whichever is longer);
12. Have a history of allergic reactions to any of the components of the investigational drug, or have a significant history of allergies to biologics;
13. Select individuals who have received or plan to receive live or attenuated vaccines within the 30 days prior to the study period;
14. Within 90 days prior to screening, blood donation or loss (excluding the amount of blood drawn during screening) exceeds 200mL;
15. Pregnant women, women planning to become pregnant during the study period, or women who are currently breastfeeding;
16. Possess fertility and refuse to use effective contraceptive methods during the trial period and within 12 weeks after the last use of medication;
17. The patients identified by the Investigators have other circumstances that make them unsuitable for participation in this study.

MAD exclusion criteria:

1. Patients with previously diagnosed diabetes (including type 1 or type 2 diabetes, etc.);
2. Start treatment with any hypoglycemic drugs within 3 months before screening;
3. Unexplained hypoglycemic events (blood sugar ≤3.9mmol/L) occurred within 1 month before screening;
4. Significant cardiovascular and cerebrovascular history within 6 months prior to screening, defined as:

   1. A history of myocardial infarction, unstable angina pectoris, coronary angioplasty or bypass surgery, valvular heart disease or heart valve repair, clinically significant arrhythmias, transient ischemic attacks, or cerebrovascular accidents; or
   2. congestive Heart failure rated III or IV by the New York Heart Association (NYHA); or
   3. The presence of ECG abnormalities (except stable coronary heart disease) that the investigator believes will affect the safety of the trial or require medical intervention;
5. History of acute or chronic pancreatitis, history of gallbladder with symptoms, history of pancreatic injury and other high-risk factors that may lead to pancreatitis;
6. Clinically significant gastric emptying abnormalities, severe chronic gastrointestinal diseases;
7. A history of depression, suicidal tendencies or behaviors, or a history of other mental illness with a clear diagnosis;
8. Have a history of organ transplantation or other acquired or congenital immune system diseases;
9. Any clinically significant endocrine system diseases;
10. Use of GLP-1 receptor (GLP-1R) agonists or GLP-1R/GCGR agonists or GIPR/GLP-1R/GCGR agonists within 3 months prior to screening;
11. Use of drugs that have an impact on body weight in the 3 months prior to screening;
12. Medullary C-cell thyroid carcinoma, multiple endocrine tumors (MEN) 2A or 2B syndrome history or family history;
13. Any type of malignancy (cured or not) within 5 years prior to screening, except cured local skin basal cell carcinoma;
14. Had undergone weight loss surgery (other than acupuncture for weight loss and local liposuction) within 1 year prior to screening, or planned to undergo any weight loss surgery or other weight loss treatment during the study period;
15. Patients with a history of severe trauma, serious infection or major surgery within 1 month before screening were judged not to be eligible for this study;
16. The results of the physical examination or laboratory examination at the time of screening meet any of the following criteria:

    1. Resting blood pressure: SBP≥160mmHg or < 90mmHg, and/or DBP≥100mmHg or < 60mmHg (one retest is allowed after 10 minutes), or addition/change of antihypertensive drugs or adjustment of antihypertensive drug dosage within 4 weeks prior to screening;
    2. Heart rate > 100 beats/min or < 50 beats/min during screening (retest once after 10 minutes is allowed);
    3. Positive for hepatitis B surface antigen (HBsAg), or positive for syphilis antibodies, or positive for human immunodeficiency virus (HIV) antibodies, or positive for hepatitis C virus (HCV) antibodies at screening;
    4. Hemoglobin abnormal;
    5. calcitonin ≥20ng/L;
    6. Hemoglobin a1C ≥6.5%;
    7. Abnormal thyroid function;
    8. Positive serum pregnancy test at screening;
    9. Liver function abnormal;
    10. Pancreatic function abnormal;
    11. Renal function abnormal;
    12. Fasting triglyceride ≥5.64mmol/L (500mg/dL), or addition/change of lipid-lowering drugs or adjustment of lipid-lowering drug dose within 4 weeks prior to screening;
17. Those who have a history of drug abuse or drug dependence within 1 year before screening;
18. There was a history of alcoholism within 1 year before screening, or regular drinking within 6 months before screening;
19. Those who have used any investigational drug or are conducting other clinical trials within the 3 months prior to screening, or whose investigational drug is within 5 half-lives (whichever is older);
20. Have a history of allergic reaction to any of the components of the investigational drug, or have a history of significant allergy to biologics;
21. Persons who have received live or attenuated vaccines within 30 days prior to screening or plan to receive live or attenuated vaccines during the study period;
22. Blood donation or blood loss (excluding blood drawn during screening) within 90 days prior to screening;
23. Pregnant women, women planning pregnancy during the study period, or women who are breastfeeding;
24. Is fertile and refuses to use effective contraceptive methods during the trial and for 12 weeks after the last dose;
25. The patients judged by the investigator had other conditions that were not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The safety of CPX101 | Up to 84 days after administration
  All AE/SAEs and other findings from vital signs(temperature, pulse, respiration, blood pressure）, physical examination(general conditions, skin, head and neck, chest, abdomen, back, four limbs, nervous system), lab tests(such as FSH, hematology, urinalysis, liver and kidney functions, electrolytes, fasting plasma glucose, blood lipids, blood amylase and lipase, calcitonin, thyroid function et al) and ECG(heart rate and measures PR, QRS, QT, and QTc intervals) will be collected from the start of screening visit to the end of the study in healthy participants
The tolerability of CPX101 | Up to 84 days after administration
  All AE/SAEs and other findings from vital signs(temperature, pulse, respiration, blood pressure）, physical examination(general conditions, skin, head and neck, chest, abdomen, back, four limbs, nervous system), lab tests(such as FSH, hematology, urinalysis, liver and kidney functions, electrolytes, fasting plasma glucose, blood lipids, blood amylase and lipase, calcitonin, thyroid function et al) and ECG(heart rate and measures PR, QRS, QT, and QTc intervals) will be collected from the start of screening visit to the end of the study in healthy participants
The safety of CPX101 | Up to 196 days after administration
  All AE/SAEs and other findings from vital signs(temperature, pulse, respiration, blood pressure）, physical examination(general conditions, skin, head and neck, chest, abdomen, back, four limbs, nervous system), lab tests(such as FSH, hematology, urinalysis, liver and kidney functions, electrolytes, fasting plasma glucose, blood lipids, blood amylase and lipase, calcitonin, thyroid function et al) and ECG(heart rate and measures PR, QRS, QT, and QTc intervals) will be collected from the start of screening visit to the end of the study in overweight and obese patients
The tolerability of CPX101 | Up to 196 days after administration
  All AE/SAEs and other findings from vital signs(temperature, pulse, respiration, blood pressure）, physical examination(general conditions, skin, head and neck, chest, abdomen, back, four limbs, nervous system), lab tests(such as FSH, hematology, urinalysis, liver and kidney functions, electrolytes, fasting plasma glucose, blood lipids, blood amylase and lipase, calcitonin, thyroid function et al) and ECG(heart rate and measures PR, QRS, QT, and QTc intervals) will be collected from the start of screening visit to the end of the study in overweight and obese patients

SECONDARY OUTCOMES:
Pharmacokinetic (PK) characteristics of CPX101 | Up to 84 days after administration
  Measurement of the concentration of CPX101 in serum after single dose injection in healthy participants
Preliminary efficacy of CPX101 | At week 16 after administration
  Evaluate the preliminary efficacy parameters (including body weight loss, waist circumference, BMI et al.) of multiple administration of CPX101 in overweight and obese patients. 1) body weight record the value in kilograms. 2) waist and hip circumference record the value in cm, Waist-to-hip ratio = waist circumference/hip circumference. 3) BMI = weight (kg) / (height [m])^2.
Pharmacokinetic (PK) characteristics of CPX101 | Up to 196 days after administration
  Measurement of the concentration of CPX101 in serum after multiple administration of CPX101 in overweight and obese patients
Immunogenicity of CPX101 | Up to 196 days after administration
  Measurement of the anti-CPX101 antibody in serum after multiple administrations in overweight and obese patients

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing hospital, Beijing, Beijing Municipality
  - Beijing Luhe hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided